CLINICAL TRIAL: NCT02319473
Title: Jakarta Acute Coronary Syndrome Registry
Acronym: JAC Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cardiovascular Center Harapan Kita Hospital Indonesia (Other)
Responsible Party: Principal Investigator, Surya Dharma, MD, PhD, Jakarta Acute Coronary Syndrome Registry, National Cardiovascular Center Harapan Kita Hospital Indonesia
Other Study IDs: JAC2007
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2017-05-05 (Actual); Status verified 2017-05

CONDITIONS: Acute Coronary Syndrome
Keywords: system of care; acute myocardial infarction; registry; Primary PCI; Fibrinolytic therapy
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: JAC Registry — patients who received acute reperfusion therapy

SUMMARY:
Jakarta acute coronary syndrome enrolled patients with acute coronary syndrome admitted to the emergency department of all health centers in Jakarta and the surrounding area.

DETAILED DESCRIPTION:
The JAC registry is an ongoing prospective, multi center, observational study that aims to enroll ACS patients who admitted to the emergency department (ED) of all health centers in Jakarta and the surrounding area. The registry has been collecting data since 2007, and used extensively since 2014.

Currently, the JAC registry is the main source of data for measuring the performance of the STEMI network in the region, namely Jakarta Cardiovascular Care Unit Network System. The STEMI network in Jakarta has been introduced as an integral part of the government project since 2010/2011.

STEMI was diagnosed based on the typical chest pain and ST segment elevation on two or more contiguos leads. The number of primary PCI, fibrinolytic therapy and non-reperfused patients were recorded.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patients that was diagnosed based on the presence of typical chest pain and ST-segment elevation in two or more contigious leads on the initial ECG

Exclusion Criteria:

* STEMI patients that was under 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All acute coronary syndrome patients admitted to the emergency department.
Sampling Method: Non-Probability Sample
Enrollment: 28812 (Estimated)
Dates: Start 2007-01; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The number of primary PCI | 15 years
In-hospital mortality | 15 years

SECONDARY OUTCOMES:
The number of fibrinolytic therapy | 15 years
The number of non-reperfused patients | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Surya Dharma, MD, PhD, Principal Investigator — National Cardiovascular Center Harapan Kita
Locations (1):
- National Cardiovascular Center Harapan Kita, Jakarta, Indonesia

REFERENCES:
- [Background] Dharma S, Andriantoro H, Purnawan I, Dakota I, Basalamah F, Hartono B, Rasmin R, Isnanijah H, Yamin M, Wijaya IP, Pratama V, Gunarto TB, Juwana YB, Suling FR, Witjaksono AM, Lasanudin HF, Iskandarsyah K, Priatna H, Tedjasukmana P, Wahyumandradi U, Kosasih A, Budhiarti IA, Pribadi W, Wirianta J, Lubiantoro U, Pramesti R, Widowati DR, Aminda SK, Basalamah MA, Rao SV. Characteristics, treatment and in-hospital outcomes of patients with STEMI in a metropolitan area of a developing country: an initial report of the extended Jakarta Acute Coronary Syndrome registry. BMJ Open. 2016 Aug 31;6(8):e012193. doi: 10.1136/bmjopen-2016-012193. PMID 27580835
- [Background] Dharma S, Andriantoro H, Dakota I, Purnawan I, Pratama V, Isnanijah H, Yamin M, Bagus T, Hartono B, Ratnaningsih E, Suling F, Basalamah MA. Organisation of reperfusion therapy for STEMI in a developing country. Open Heart. 2015 May 21;2(1):e000240. doi: 10.1136/openhrt-2015-000240. eCollection 2015. PMID 26019883
- [Background] Dharma S, Siswanto BB, Firdaus I, Dakota I, Andriantoro H, Wardeh AJ, van der Laarse A, Jukema JW. Temporal trends of system of care for STEMI: insights from the Jakarta Cardiovascular Care Unit Network System. PLoS One. 2014 Feb 10;9(2):e86665. doi: 10.1371/journal.pone.0086665. eCollection 2014. PMID 24520322
- [Background] Dharma S, Juzar DA, Firdaus I, Soerianata S, Wardeh AJ, Jukema JW. Acute myocardial infarction system of care in the third world. Neth Heart J. 2012 Jun;20(6):254-9. doi: 10.1007/s12471-012-0259-9. PMID 22328356
- [Derived] Dharma S, Mahavira A, Haryono N, Sukmawan R, Dakota I, Siswanto BB, Rao SV. Association of Hyperglycemia and Final TIMI Flow with One-Year Mortality of Patients with Acute ST-Segment Elevation Myocardial Infarction Undergoing Primary PCI. Int J Angiol. 2019 Sep;28(3):182-187. doi: 10.1055/s-0039-1691811. Epub 2019 Jun 17. PMID 31452586